CLINICAL TRIAL: NCT05811546
Title: Immunohistochemical Evaluation of DNA Methylation and Histone Modification in H. Pylori Associated Gastric Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliyah Soliman Ali, Pathology resident, Assiut University
Other Study IDs: Epigenetics Gastric Carcinoma
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Formalin-fixed-paraffin-embedded tissue specimens.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- H. pylori Gastritis specimens
  Interventions: Diagnostic Test: Immunohistochemical staining for DNMT1 and EZH2
- Non-H. pylori Gastritis specimens
- Gastric carcinoma specimens

INTERVENTIONS:
Diagnostic Test: Immunohistochemical staining for DNMT1 and EZH2 — Immunohistochemical staining for DNMT1 and EZH2 using rabbit monoclonal/polycolonal antibodies with immunoperoxidase staining will be used as a visualization method. Antibodies dilutions, antigen retrieval methods, and incubation time will all be conducted according to the manufacturer's instructions.
  Groups: H. pylori Gastritis specimens

SUMMARY:
The goal of this cross-sectional study is to evaluate epigenetic modifications in gastric carcinogenesis, mainly in H. pylori gastritis vs gastric carcinoma. The main question[s] it aims to answer are:

* How does H. pylori infection cause gastric cancer?
* Can DNA methylation and other epigenetic changes predict and affect the development of gastric cancer? Formalin-fixed-paraffin-embedded tissue specimens will be obtained and reviewed for comparison between epigenetic changes in H. pylori gastritis and gastric adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Resected specimens and endoscopic guided biopsies of intestinal type gastric carcinoma, H. Pylori associated gastritis, and non-H. Pylori gastritis with:
* Available full clinical data: (age, sex, complaint, findings in clinical examination).
* Full data of previous endoscopy and radiology.

Exclusion Criteria:

* Cases of diffuse type gastric carcinoma.
* Any case of gastric cancer, H. Pylori associated gastritis, non-H. Pylori gastritis, benign gastric lesions with missing clinical, endoscopic, radiologic or follow-up data.
* Cases with no available H&E stained slides or formalin fixed paraffin embedded block.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Formalin-fixed-paraffin-embedded tissue blocks from resected specimens and endoscopic guided biopsies of intestinal type gastric carcinoma, H. Pylori associated gastritis, and non-H. Pylori gastritis.
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in DNMT1 and EZH2 expression. | two years
  Histopathological evaluation of routine H&E slides and immunohistochemical markers to compare the intensity and extent of epigenetic changes in both H. Pylori associated gastritis and gastric carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No